CLINICAL TRIAL: NCT05666518
Title: Vericiguat Drug Use Two-arm Investigation in Chronic Heart Failure
Brief Title: A Study to Learn More About the Safety of the Drug Vericiguat in Japanese People With Chronic Heart Failure Who Will be Receiving Vericiguat Under Real-world Conditions
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21880
Record Dates: First submitted 2022-12-02; First posted 2022-12-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — vericiguat; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vericiguat arm: Japanese patients with a diagnosis of chronic heart failure who received standard treatment and will start vericiguat therapy for chronic heart failure.
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)
- control arm: Japanese patients a diagnosis of chronic heart failure who received standard treatment and will continue standard of care treatment for chronic heart failure.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Dosage at the discretion of the treating physician, based on the recommendations written in the product information.
  Groups: vericiguat arm
Drug: Standard of care — Dosage at the discretion of the treating physician
  Groups: control arm

SUMMARY:
This is an observational study in which data from Japanese people with chronic heart failure who will be receiving vericiguat is studied.

Chronic heart failure (HF) is a long-term condition where the heart does not pump blood as well as it should. Heart failure can lead to other serious medical conditions, and it can lead to hospitalization or death.

The drug vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC). The sGC enzyme helps regulate the heart and blood circulation. Vericiguat is already available and approved for doctors to prescribe to people who have heart failure. A limited number of patients have been treated with vericiguat. Therefore information about its safety in a broader population and especially among Japanese people as well as for prolonged periods of treatment is still missing.

In this study, the researchers want to learn more about how safe vericiguat is if used in Japanese people with long term HF. To see how safe vericiguat is, the researchers will collect the medical problems the participants have during the treatment with vericiguat under real-word conditions. They will particularly focus on the following:

* high blood pressure
* any medical problems due to combination of the study treatment vericiguat with nitrates and nitric oxide (NO) donors or with PDE5 inhibitors
* medical problems in participants with liver problems or with reduced kidney function
* medical problems in participants with low blood pressure below <100 mmHg or with symptoms due to low blood pressure
* any medical problems after prolonged periods of treatment with vericiguat. These medical problems are also known as "adverse events" (AEs) which may or may not be related to the study treatment.

In addition, this study will gather information about how long vericiguat treatment can prevent death caused by cardiovascular problems such as heart attack and stroke compared to standard of care. Cardiovascular death (safety specification) will be assessed in a comparative manner with the control arm as the primary objective

The participants will receive their treatments as prescribed by their doctors according to the approved product information. The data for this study will be collected using an electronic case report form (eCRF) and medical records. The following data from the study participants will be documented during visits that take place in routine practice:

* underlying and concomitant diseases,
* prior medication,
* treatment duration,
* laboratory parameters,
* vital signs,
* results of cardiac exams (e.g. cardiac ultrasound),
* heart failure related hospitalization events,
* adverse events. The data collection will start from the beginning of vericiguat/standard of care treatment and will cover a time period of 2 years unless no further information can be expected from the participant at a given point in time, or death.

The total study duration will be six years, including data analysis and cleaning.

ELIGIBILITY:
Inclusion Criteria:

vericiguat arm:

* Patients receiving standard treatment for chronic heart failure, and vericiguat will be treated in accordance with the package insert (no history of receiving vericiguat)
* Patients who gave written consent to this investigation

control arm:

* Patients receiving standard treatment for chronic heart failure according to the package insert of vericiguat as following (no history of receiving vericiguat)

  * Prior (within 6 months) heart failure hospitalization or prior (within 3 months) intravenous (IV) diuretics for heart failure not requiring hospitalization (This will be applied only for the first ~75% of patients meeting this criteria to be enrolled.) Note: No more than approximately 25% of patients without a qualifying history of prior heart failure hospitalization within 6 months or prior IV diuretics for heart failure not requiring hospitalization within 3 months can be enrolled in the study.
  * New York Heart Association (NYHA) Classification: Class II to Class IV
  * Left ventricular ejection fraction (LVEF): less than 45%
* Patients who gave written informed consent to this study

Exclusion Criteria:

vericiguat arm:

- Patients who are participating in an interventional study

control arm:

* Patients who have started or are scheduled to start therapy with vericiguat for chronic heart failure
* Patients who are participating in an interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of Japanese patients with chronic heart failure have been prescribed vericiguat or standard treatment by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of Adverse Events (AEs) for vericiguat arm | Up to 2 years.
Seriousness of Adverse Events (AEs) for vericiguat arm | Up to 2 years
Outcome of Adverse Events (AEs) for vericiguat arm | Up to 2 years
Causality assessment of Adverse Events (AEs) for vericiguat arm | Up to 2 years
Incidence of Cardiovascular (CV) death for vericiguat arm and control arm | Up to 2 years
  Definition of CV death is Heart failure, acute myocardial infarction, stroke (cerebral infarction, cerebral hemorrhage), sudden death, other CV deaths (e.g., pulmonary embolism, peripheral arterial disease), death of unknown cause

SECONDARY OUTCOMES:
The duration (days) of vericiguat treatment for vericiguat arm | Up to 2 years
The reason for ending vericiguat treatment/observation for vericiguat arm | Up to 2 years
Dosage and dose modification of vericiguat treatment for vericiguat arm | Up to 2 years
Systolic blood pressure and diastolic blood pressure for vericiguat arm | Up to 2 years
Pulse rate for vericiguat arm | Up to 2 years
Assessment of left ventricular end-diastolic volume index and left ventricular end-systolic volume index for vericiguat arm | Up to 2 years
Assessment of left ventricular ejection fraction for vericiguat arm | Up to 2 years
Assessment of Brain Natriuretic Peptide/N-terminal pro-Brain Natriuretic Peptide for vericiguat arm | Up to 2 years
Assessment of Serum creatinine for vericiguat arm | Up to 2 years
Assessment of e-GFR for vericiguat arm | Up to 2 years
Assessment of Hemoglobin for vericiguat arm | Up to 2 years
Assessment of Hematocrit for vericiguat arm | Up to 2 years
Assessment of New York Heart Association (NYHA) classification for vericiguat arm | Up to 2 years
Concomitant medications for vericiguat arm | Up to 2 years
All-cause mortality for vericiguat arm | Up to 2 years
Number of patients with Heart Failure (HF) hospitalization during observation period for vericiguat arm | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Japanese registries, Multiple Locations, Many Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.